CLINICAL TRIAL: NCT02932553
Title: BVS Implantation in Patients With Variant Angina and MODerate Coronary Artery Disease: Pilot Study
Brief Title: BVS Implantation in Patients With Variant Angina and MODerate Coronary Artery Disease
Acronym: BIVA-pilot
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: BVS was withdrawn from the market
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, professor, Division of Cardiology, Department of Internal Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2016-22
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Angina Pectoris, Variant
Keywords: bioresorbable vascular scaffold; variant angina; moderate coronary artery disease; vasospastic angina
MeSH Terms: conditions — Angina Pectoris, Variant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BVS and OMT (Experimental): Optimal medical treatment + BVS implantation
  Interventions: Device: BVS+OMT

INTERVENTIONS:
Device: BVS+OMT — bioresorbable vascular scaffold implantation plus optimal medical treatment

SUMMARY:
The purpose of this study is to determine whether BVS(Bioresorbable Vascular Scaffold) implantation with optimal medical therapy can improve the outcome of patients with variant angina and moderate coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and more
* Vasospastic angina diagnosed by provocation test including ergonovine provocation coronary angiography or ergonovine echocardiogram
* No-ischemia producing moderate coronary artery disease(stenosis>50%, FFR>0.8)

Exclusion Criteria:

* Ischemic coronary lesion
* Organic heart disease associated with myocardial ischemia or sudden cardiac death
* History of percutaneous coronary intervention
* Cerebrovascular diseases or peripheral disease
* NYHA III and IV
* Cardiac pacemaker or implantable defibrillator
* Pregnancy or breast feeding
* Life expectancy less than 2 years

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-19 (Actual)

PRIMARY OUTCOMES:
Composite of all cause death, myocardial infarction, and angina-related hospitalization | 2year

SECONDARY OUTCOMES:
Variant angina | 2year
  by Ergonovine test
All cause death | 2year
Cardiac death | 2year
Repeat revascularization | 2year
Scaffold thrombosis | 2year
Myocardial infarction | 2year
Stroke | 2year
Angina-related hospitalization | 2year
Composite event of death or myocardial infarction | 2year
Composite event of cardiac death or myocardial infarction | 2year

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided